CLINICAL TRIAL: NCT04281121
Title: the Effect of Omega 3 Fatty Acids Supplements on Antioxidant Capacity in Egyptian Children With Non Alcoholic Fatty Liver Disease
Brief Title: Omega 3 Supplementation in Children With Non Alcoholic Fatty Liver
Acronym: omega 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, yasmin gamal el gendy, professor of pediatrics, Ain Shams University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD 44/2017
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- supplemented (Active Comparator): Life style modification, diet regimen and Omega-3 fatty acids supplementation
  Interventions: Dietary Supplement: omega 3 fatty acids
- non supplemented (Active Comparator): Life style modification and diet regimen
  Interventions: Dietary Supplement: omega 3 fatty acids

INTERVENTIONS:
Dietary Supplement: omega 3 fatty acids — : Life style modification, diet regimen and Omega-3 fatty acids supplementation: The dose of omega-3 fatty acids depended on the weight of patients according to World Health Organization recommendations 400 milligrams per 10 kilograms of body weight and had been given into two doses per day, before morning and evening meals

SUMMARY:
this is a prospective, interventional, open-label, randomized study on the efficacy of omega 3 fatty acids supplementation in Egyptian children with non-alcoholic fatty liver disease who had been selected from nutrition and outpatient clinic at Pediatric hospital, Ain Shams University

ELIGIBILITY:
Inclusion Criteria:

Children between 5 - 16 years old with diffusely hyper echogenic liver at ultrasonography were included in the study.

Exclusion Criteria:

* Patients with secondary causes of steatosis including total parenteral nutrition, drugs causing fatty liver disease for example steroids, hepatitis A, B, C, cytomegalovirus, Epstein-Barr virus infections, autoimmune liver disease, metabolic liver diseases, Wilson's disease, and alpha-1-antitrypsin deficiency.
* Patients currently taking fish oil supplements.
* Patients with systemic illness such as cardiac and kidney diseases.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
grade of fatty liver in children | 3 month
  improvement

CONTACTS AND LOCATIONS:
Overall Officials: zeinab Kabbany, professor, Principal Investigator — Ain Shmas University
Locations (1):
- Pediatrics hospital Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No